CLINICAL TRIAL: NCT00282230
Title: A Phase 2, Randomized, Open-Label, Parallel Group, Multi-Center Study to Assess the Safety and Efficacy of Prograf®/FK778 and Prograf®/MMF in De Novo Kidney Transplant Recipients
Brief Title: A Study to Evaluate the Safety and Efficacy of Prograf/FK778 and Prograf/MMF in de Novo Kidney Transplant Recipients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma US, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03-0-165
Record Dates: First submitted 2006-01-24; First posted 2006-01-26 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2012-06

CONDITIONS: Kidney Transplantation
Keywords: Malononitrilamide; immunosuppression; treatment efficacy; treatment outcome
MeSH Terms: interventions — 2-cyano-3-hydroxy-N-(4-(trifluoromethyl)phenyl)-2-hepten-6-ynamide

INTERVENTIONS:
Drug: FK778

SUMMARY:
A study to evaluate the safety and efficacy of Prograf/FK778 in de novo kidney transplant patients

ELIGIBILITY:
Inclusion Criteria:

* Patient is a recipient of a primary or retransplanted cadaveric or non-HLA-identical living donor kidney.
* Patient must receive first oral dose of randomized study drug within 48 hours of transplant procedure.

Exclusion Criteria:

* Patient has received or is receiving an organ transplant other than kidney
* Patient has received a kidney transplant from a cadaveric donor >= 60 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2003-11; Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Incidence of biopsy confirmed acute rejection (Banff Grade ≥ I) at 6 months.

SECONDARY OUTCOMES:
6 month patient and graft survival rates
time to first biopsy confirmed acute rejection
clinically treated acute rejection episodes
treatment failure (up to 6 months)
renal function (SrCl and CrCl)
quantitation of CMV and polyomavirus viral load

CONTACTS AND LOCATIONS:
Overall Officials: John Holman, MD, Study Director — Astellas Pharma US, Inc.
Locations (22):
- United States (22):
  - Birmingham, Alabama
  - Los Angeles, California
  - San Diego, California
  - Denver, Colorado
  - Washington D.C., District of Columbia
  - Jacksonville, Florida
  - Miami, Florida
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Wichita, Kansas
  - New Orleans, Louisiana
  - Detroit, Michigan
  - New Brunswick, New Jersey
  - New York, New York
  - Durham, North Carolina
  - Cincinnati, Ohio
  - Harrisburg, Pennsylvania
  - Philadelphia, Pennsylvania
  - Memphis, Tennessee
  - Salt Lake City, Utah
  - Madison, Wisconsin
  - Milwaukee, Wisconsin